CLINICAL TRIAL: NCT00501397
Title: An Open Label Study in Healthy Volunteers to Investigate the Effect of Ketoconazole on the Pharmacokinetics of GSK189075
Brief Title: A Study of the Effects of Ketoconazole Taken Orally Has on the PK Profiles of a Dose of GSK189075 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KG2108197
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: ketoconazole,; drug interaction,; pharmacokinetics; T2DM,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ketoconazole
Drug: GSK189075
  Other Names: ketoconazole

SUMMARY:
The purpose of this research study is to evaluate the effect of several daily doses of ketoconazole (a medication used to treat fungal infections like athlete's foot) on a single dose of GSK189075 (an experimental diabetes drug), and also to evaluate the safety and tolerability of GSK189075 in healthy volunteers. The study will see whether ketoconazole causes GSK189075 to stay in your bloodstream for a longer period of time. It will also examine whether GSK189075 causes any changes in the amount of glucose you have in your urine.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy, non-smoking male or female.
* Are 18 to 55 years old, inclusive.
* Have a body weight of > or equal to 110 pounds.
* Are a female who is unable to have any more children and have a negative pregnancy test.
* Are willing and able to provide written informed consent before the start of any study-related procedures.
* Are able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions.

Exclusion Criteria:

* Smoke or use any tobacco products.
* Have a known allergic reaction to ketoconazole or study drug.
* Have a history of regular alcohol consumption greater than 7 drinks per week for females or greater than 14 drinks per week for males.
* Have a positive drug or alcohol or smoking test at screening or check-in to the clinic.
* Have participated in another clinical trial within 30 days prior to screening in which you have received an investigational drug.
* Have donated a pint of blood within 56 days before the first dose of study drug.
* Have any known or suspected stomach condition (or stomach surgery within the 6 months prior to dosing).
* Have abnormal liver test results.
* Have a documented history or diagnosis of cirrhosis.
* Have positive results for hepatitis C or B, or HIV at screening.
* Have blood pressure outside of the normal range.
* Are a male subject who is unwilling to either abstain from sexual activity or unwilling to use birth control during the course of the study.
* Are using non-prescription drugs, vitamins, herbal or dietary supplements (including St John's Wort) within 7 days before the first dose of study medication,
* Have any abnormality identified on the screening physical or laboratory examination that the study physician feels would make it inappropriate for you to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Plasma blood samples for GSK189075 at Day 1 Session 1, Days 5 & 6 Session 3 | at Day 1 Session 1, Days 5 & 6 Session 3 urine collections for volume
urine collections for volume, glucose, & creatinine at Day 1 Session 1, Days 5 & 6 Session 3. | at Day 1 Session 1, Days 5 & 6 Session 3.

SECONDARY OUTCOMES:
Adverse events: all visits | all visits
ECG,labs: Screening,Days -1 & 1 Session 1,Day 4 Session 2,Days 5-6 Session 3 | Screening,Days -1 & 1 Session 1,Day 4 Session 2,Days 5-6 Session 3
Labs:followup | followup
Urine: Day 1 Session 1,Days 5-6 Session 3 | Day 1 Session 1,Days 5-6 Session 3
Vitals: Screening,Days -1 & 1 Session 1,Days 1-4 Session 2,Days 5-6 Session 3,followup | Screening,Days -1 & 1 Session 1,Days 1-4 Session 2,Days 5-6 Session 3,followup

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Columbus, Ohio, United States